CLINICAL TRIAL: NCT04752345
Title: A Prospective Randomized Multi-center Clinical Trial Comparing Different Fibrinolysis-transfer Percutaneous Coronary Intervention Strategies in Acute ST-segment Elevation Myocardial Infarction
Brief Title: Optimal Reperfusion Strategy for STEMI Patients With Anticipated PPCI Delay
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yong He, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WestChinaH-CVD-002
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-01

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: ST-elevation myocardial infarction; primary percutaneous coronary; pharmacoinvasive strategy; reduced-dose fibrinolysis
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Pharmacoinvasive strategy, fibrinolysis combined with rescue PCI (in case of failed fibrinolysis) or routine early invasive strategy (in case of successful fibrinolysis)
  Interventions: Other: Pharmacoinvasive strategy
- Experimental group (Experimental): Reduced-dose fibrinolysis combined with immediate invasive therapy
  Interventions: Other: Reduced-dose facilitated PCI strategy

INTERVENTIONS:
Other: Pharmacoinvasive strategy — Pharmacoinvasive treatment [full-dose fibrinolysis combined with rescue PCI (in case of failed fibrinolysis) or routine early PCI (3 to 24 hours, in case of successful fibrinolysis)
  Arms: Control group
Other: Reduced-dose facilitated PCI strategy — Reduced-dose facilitated PCI[reduced-dose fibrinolysis,simultaneously transfer,immediate coronary angiography and andioplasty when arrived at PCI center(<3 hours)]
  Arms: Experimental group

SUMMARY:
The OPTIMAL-REPERFUSION trial will help determine whether reduced-dose facilitated PCI strategy improves clinical outcomes in patients with STEMI and anticipated PPCI delay

DETAILED DESCRIPTION:
OPTIMAL-REPERFUSION is an investigator-initiated, prospective, multicenter, randomized, open-label, superiority trial with blinded evaluation of outcomes. A total of 632 STEMI patients presenting within 6 hours after symptom onset and with an expected time of medical contact to percutaneous coronary intervention ≥120 min will be randomized to a reduced-dose facilitated PCI strategy (reduced-dose fibrinolysis combined with simultaneous transfer for immediate invasive therapy with a time interval between fibrinolysis to PCI < 3 hours) or to pharmacoinvasive treatment. The primary endpoint is the composite of death, reinfarction, refractory ischemia, congestive heart failure, or cardiogenic shock at 30-days.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over and less than 75 years old;
* Patents with STEMI with symptom onset persisted more than 30mim and within 6 h before randomization;
* ECG >=2 mm ST-segment elevation in 2 contiguous precordial leads or >=1 mm ST- segment elevation in 2 contiguous extremity leads, or new left bundle branch block;
* Patents with an expected time from FMC to PCI >=120 min.
* Signed informed consent form prior to trial participation.

Exclusion Criteria:

* Fibrinolysis contradictions: Definite hemorrhagic stroke history;ischemic stroke or cerebrovascular accident in nearly 6 months;
* Any history of central nervous system damage (i.e. neoplasm, aneurysm, intracranial or spinal surgery) or recent trauma to the head or cranium (i.e. < 3 months);
* Active bleeding or known bleeding disorder/diathesis; Recent administration of any i.v. or s.c. anticoagulation within 12 hours including unfractionated heparin, enoxaparin and/or bivalirudin or current use of oral anticoagulation (warfarin or coumadin);
* Arterial aneurysm, arterial/venous malformation and aorta dissection; Uncontrolled hypertension, defined as a single blood pressure measurement >=180/110 mm Hg (systolic BP >=180 mm Hg and/or diastolic BP >=110 mm Hg) prior to randomisation;
* Major surgery, biopsy of a parenchymal organ, noncompressible vascular puncture, or significant trauma within the past 2 months (this includes any trauma associated with the current myocardial infarction);
* prolonged or traumatic cardiopulmonary resuscitation (> 10 minutes) within the past 2 weeks; major surgery pending in the following 30 days. 2. Complex heart condition Evidence of cardiac rupture; Pre-existing heart failure and previous New York heart function classification III-IVCardiogenic shock (SBP <90mmHg after fluid infusion or SBP<100mmHg after vasoactive drugs);
* PCI within previous 1 month or previous bypass surgery;
* Myocardial infarction in the past year or previously known coronary artery disease not suitable for revascularization;
* Known acute pericarditis and/or subacute bacterial endocarditis;
* Hospitalization for cardiac reason within past 48 hours;
* Severe comorbidity: Other diseases with life expectancy <=12 months;
* Any history of severe renal or hepatic dysfunction (hepatic failure, cirrhosis, portal hypertension or active hepatitis);
* neutropenia, thrombocytopenia;
* Severe COPD with hypoxemia;
* Not suitable for clinical trial: Inclusion in another clinical trial; Previous enrollment in this study or treatment with an investigational drug or device under another study protocol in the past 7 days;
* Pregnant or lactating;
* Body weight <40kg;
* Known hypersensitivity to any drug that may be used in the study;
* Inability to follow the protocol and comply with follow-up requirements or any other reason the investigator feels would place the patient at increased risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 632 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
The rate of major composite endpoint events | 30 days
  Composite of death, reinfarction, refractory ischaemia, congestive heart failure, or cardiogenic shock

SECONDARY OUTCOMES:
The rate of major ventricular arrhythmia | 1 year
  Ventricular arrhythmias, occurring more than 6 hours after randomization, persisting for at least 30 seconds, and accompanying with unstable hemodynamics that required electrical cardioversion / defibrillation
The rate of ischemia stroke | 1 year
  Defined as the presence of a new focal neurologic deficit thought to be vascular in origin, with signs or symptoms lasting more than 24 hours. It is strongly recommended (but not required) that an imaging procedure such as a computerized tomography (CT) or magnetic resonance imaging (MRI) be performed.
The rate of death | 1 year
  Death will be classified as cardiovascular or non-cardiovascular.
The rate of reinfarction | 1 year
  Recurrent symptoms or signs of cardiac ischemia lasting more than 30 minutes with new ST-T segment changes or Q-wave in at least 2 contiguous leads or new onset LBBB and recurrent significant increase in cardiac enzyme levels. The increase in CK-MB level is considered significant when it occurs after at least a ≥25% decrease in CK-MB from a prior peak level and is >2 times the upper limit of normal (ULN) in the absence of coronary interventions, or >5 times above the ULN after PCI
The rate of stent thrombosis | 1 year
  The stent thrombosis are defined in accordance with the Academic Research Consortium (ARC) definitions
The rate of target vessel revascularization | 1year
  The target vessel revascularizationare defined in accordance with the Academic Research Consortium (ARC) definitions
The rate of congestive heart failure | 1 year
  New or worsening congestive heart failure will be considered as patients presenting with at least one of the following conditions and requiring treatment with diuretics: 1) Pulmonary oedema/congestion on chest X-ray without suspicion of a non-cardiac cause; 2) Rales >1/3 up from the lung base; 3) Pulmonary capillary wedge pressure (PCWP) >25 mmHg; 4) Dyspnea with PO2 < 80 mmHg or O2 sat < 90 % (no supplemental O2) in the absence of known lung disease.
The rate of Cardiogenic shock | 1 year
  The manifestation of vascular collapse and shock (systolic BP < 90 mmHg for at least 30 min or systolic BP > 90 mmHg after inotropic or intra-aortic balloon support with a cardiac index < 2.2 L/min/m2 or < 2.5 L/min/m2 after inotropic or intra-aortic balloon support, peripheral signs of hypoperfusion, and chest X-ray with pulmonary edema
Number of Participants with TIMI flow grade (TFG) 3 for epicardial reperfusion | 1 minute after stent was deployed
  TIMI flow grade (TFG) 3 for epicardial reperfusion
Number of Participants with TIMI myocardial perfusion grade (TMPG) 3 for myocardial reperfusion | 1 minute after stent was deployed
  TIMI myocardial perfusion grade (TMPG) 3 for myocardial reperfusion
Resolution of the initial sum of ST- segment elevation (STR) ≥ 70% post catheterization | 60min after the stent was deployed
  Resolution of the initial sum of ST- segment elevation (STR) ≥ 70% post catheterization
Peak CK-MB level | 48 hours after system onset
  Peak CK-MB level
Adverse events | 1 year
  Intracranial bleeding or major bleeding

OTHER OUTCOMES:
Cost-effectiveness of reduced-dose pharmacoinvasive strategy compared to current care | 1 year
  The total costs during the first 12 months include resources used during the first hospitalization including transportation and catheterization procedures, medications, examinations, management of complications and subsequent hospital admissions for cardiovascular problems in the first year after STEMI
Health-related quality of life | 1 year
  Measured with EQ-5D questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Yong He, Principal Investigator — Department of Cardiology, West China Hospital of Sichuan University

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared within six months after the trial finished through Electronic data capture system or ResMan
Supporting Information: Study Protocol
Time Frame: Within six months after the trial complete

REFERENCES:
- [Derived] Chen Z, Wang D, Ma M, Li C, Wan Z, Zhang L, Zhu Y, Wang M, Wang H, He S, Peng Y, Wei J, Huang B, He Y; OPTIMAL-REPERFUSION trial investigator. Rationale and design of the OPTIMAL-REPERFUSION trial: A prospective randomized multi-center clinical trial comparing different fibrinolysis-transfer percutaneous coronary intervention strategies in acute ST-segment elevation myocardial infarction. Clin Cardiol. 2021 Apr;44(4):455-462. doi: 10.1002/clc.23582. Epub 2021 Feb 25. PMID 33634478